CLINICAL TRIAL: NCT00004242
Title: Phase I Study of Oxaliplatin in Combination With 5-Fluorouracil and Gemcitabine in Patients With Solid Tumors
Brief Title: Combination Chemotherapy in Treating Patients With Metastatic or Unresectable Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067487; AECM-1199904138; NCI-T99-0023; NYU-9944
Record Dates: First submitted 2000-01-28; First posted 2003-12-11 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2002-07

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Fluorouracil; Gemcitabine; Oxaliplatin

ARMS (1):
- Arm I (Experimental): See detailed description.
  Interventions: Drug: fluorouracil; Drug: gemcitabine hydrochloride; Drug: oxaliplatin

INTERVENTIONS:
Drug: fluorouracil
Drug: gemcitabine hydrochloride
Drug: oxaliplatin

SUMMARY:
Phase I trial to study the effectiveness of combination chemotherapy in treating patients who have metastatic or unresectable solid tumors. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose, recommended phase II dose, and associated toxic effects of the triple combination of continuous infusion fluorouracil, weekly gemcitabine, and oxaliplatin in patients with metastatic or unresectable solid tumors.

II. Define sequence dependent toxic effects, if any, and establish pharmacokinetic and pharmacodynamic relationships in context of this triple combination chemotherapy in this patient population.

OUTLINE: This is a dose-escalation study of oxaliplatin and gemcitabine.

For course 1, and then course 3 and beyond, patients receive oxaliplatin IV over 2 hours on day 1, followed by gemcitabine IV over 30 minutes on days 1 and 8, and then fluorouracil IV continuously on days 1-14. For course 2, patients receive treatment in the same manner as in course 1, except gemcitabine is given initially, followed by oxaliplatin, and then fluorouracil. Treatment continues every 21 days in the absence of unacceptable toxicity or disease progression.

Cohorts of 1-6 patients receive escalating doses of oxaliplatin and gemcitabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. The recommended phase II dose (RPTD) is defined as the dose preceding MTD.

Once RPTD is defined, the cohort is expanded to an additional 13 patients. These patients receive a fixed dose of oxaliplatin, gemcitabine, and fluorouracil as determined by the phase I dose escalation portion of this study.

Patients are followed for disease progression.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or clinically confirmed metastatic or unresectable solid tumor for which no standard curative or palliative therapy exists or is no longer
* No known brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm3
* Platelet count at least 100,000/mm3

Hepatic:

* Bilirubin normal
* Proven Gilbert's syndrome (UGT1A1 promoter mutation or clinical
* documentation of stress bilirubin levels) allowed
* AST/ALT no greater than 3 times upper limit of normal

Renal:

* Creatinine normal OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Pulmonary:

* No unexplained respiratory problems (e.g., nonproductive cough, dyspnea,
* rales, pulmonary infiltrates, hypoxia, or tachypnea)

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No clinical evidence of neuropathy
* No prior allergy to platinum compounds
* No prior allergy to antiemetics appropriate for administration in
* conjunction with protocol directed chemotherapy
* No other concurrent uncontrolled illness (e.g., active infection)

PRIOR CONCURRENT THERAPY:

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas and
* platinum) and recovered
* No more than 1 prior chemotherapy regimen for cancer

Radiotherapy:

* At least 4 weeks since prior radiotherapy

Other:

* No concurrent antiretroviral agents (HAART)
* No other concurrent investigational agents or commercial therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 1999-10; Primary Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard S. Hochster, MD, Study Chair — NYU Langone Health
Locations (2):
- United States (2):
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York

REFERENCES:
- [Result] Basu S, Goel S, Hochster H, et al.: Phase I and pharmacokinetic (PK) study of oxaliplatin (Ox) with gemcitabine (Gem) and continuous intravenous (CIV) infusion 5-fluorouracil (FU) in patients with advanced solid malignancies. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-2132, 2002.